CLINICAL TRIAL: NCT00628667
Title: A Multicenter, Double -Blind, Placebo-controlled Study to Evaluate the Effects of Esomeprazole 40mg Bid on the Signs and Symptoms of Chronic Posterior Laryngitis With Suspected Laryngopharyngeal Reflux
Brief Title: Chronic Posterior Laryngitis With Suspected Laryngopharyngeal Reflux
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD - Nexium Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH-NEE-0002; D9611C00002
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Posterior Laryngitis (CPL)
Keywords: Chronic Posterior Laryngitis; CPL; Pharyngeal acid reflux; Esomeprazole; Nexium
MeSH Terms: interventions — Esomeprazole

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Esomeprazole
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — 40mg orally twice daily
  Other Names: Nexium
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
This study looks at how effective acid suppression therapy is on symptoms associated with chronic posterior laryngitis (CPL) in patients with documented pharyngeal acid reflux.

ELIGIBILITY:
Inclusion Criteria:

* One or more of the following symptoms present for at least 3 consecutive months: throat clearing, cough, globus, sore throat, or hoarseness.
* Patients must complete a run-in diary card, and this will be looked at to ensure met the inclusion criteria.
* Must have a total score of 5 or more on the Chronic Posterior Laryngitis Index (CPLI) grading system.

Exclusion Criteria:

* A number of diseases / conditions would preclude a patient from taking part in the study, as listed in the protocol.
* If the patient is on certain medications this will also preclude them from taking part.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2002-02; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Daily diary cards and investigator symptom assessment to evaluate the efficacy of acid suppression therapy on symptoms associated with chronic posterior laryngitis (CPL) in patients without documented pharyngeal acid | Dialy diary cards, investigator assessments, laryngoscopy at week 16

SECONDARY OUTCOMES:
Daily diary cards and investigator symptom assessment throughout to evaluate the efficacy of acid suppression therapy on resolution of signs of CPL at weeks 8 and 16 in patients without documented pharyngeal acid reflux. | Dialy diary cards, investigator assessments, laryngoscopy at weeks 8 and 16
Quality of life Questionnaire | Quality of life questionnaire completed at screening and week 16
To evaluate the safety and tolerability by collecting an ongoing record of adverse events. | Ongoing to week 16.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca